CLINICAL TRIAL: NCT02868164
Title: Fecal Microbiota Therapy Versus Standard Therapy in Decompensated NASH Related Cirrhosis: A Randomized Controlled Trial.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-05
Record Dates: First submitted 2016-08-04; First posted 2016-08-16 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2018-02

CONDITIONS: NASH Related Decompensated Cirrhosis
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (FMT) (Experimental)
  Interventions: Drug: Fecal Microbiota Transplantation
- Weight Reduction (Active Comparator)
  Interventions: Drug: Standard Treatment; Other: Weight Reduction

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — The recipient will receive healthy donor, prepared fecal installations through a Naso-gastric tube, 100 ml once a month for 6 month.
  Arms: Fecal Microbiota Transplantation (FMT)
Drug: Standard Treatment — Standard Treatment
  Arms: Weight Reduction
Other: Weight Reduction — routine exercise for weight reduction
  Arms: Weight Reduction

SUMMARY:
The study will be conducted in the Department of Hepatology, Institute of Liver & Biliary Sciences, New Delhi. As a part of this study history will be taken and clinical examination will be done. Subjects will be screened for diagnosis of NASH (Non Alcoholic Steatohepatitis) cirrhosis. If subjects are found to have NASH (Non Alcoholic Steatohepatitis) cirrhosis, they will be chosen to receive stool from healthy donor, which is voluntarily donated by a healthy donor related or unrelated to the subjects and the stool will be prepared using standard guidelines. The prepared sample of stool, about 50 ml will be instilled into proximal small intestine by way of a thin and soft tube inserted through nose. This administration of sample, 50 ml daily will occur once a month every month for 6 months. The liver function parameters will be assessed and thereafter at 1 month and 3 months & subjects will be clinically assessed for improvement or worsening.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years.
2. All patients with cirrhosis with current or previous histological evidence of steatosis or steatohepatitis.
3. Histological evidence of definite or probable NASH (Non Alcoholic Steatohepatitis) based upon a liver biopsy prior to enrollment and a NAFLD (Non Alcoholic Fatty Liver Disease) activity score (NAS) ≥5 with ≥1 in each component of the NAS score (steatosis, scored 0-3, ballooning degeneration, 0-2, and lobular inflammation, 0-3).
4. No history of recent spontaneous bacterial peritonitis.(1 month)
5. Child Pugh Score of 6 - 10

Exclusion Criteria:

1. Diagnosis of liver disease other than NASH (Non Alcoholic Steatohepatitis) cirrhosis
2. Ongoing bacterial infection requiring antibiotic treatment.
3. Current or history of significant alcohol consumption for a period of more than 3
4. consecutive months within 1 year prior to screening
5. Treatment with antibiotics or probiotics in the preceding 3 months.
6. Inability to safely obtain a liver biopsy in compensated cirrhosis or to perform an upper GastroIntestinal endoscopy
7. Pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events complication rate in NASH (Non Alcoholic Steatohepatitis) patients in both groups | 1 year
  Adverse events like GastroIntestinal Bleed, development of ascites, Spontaneous Bacterial peritonitis, ACLF (acute on chronic liver failure)

SECONDARY OUTCOMES:
Reduction in HVPG (Hepatic Venous Pressure Gradient) in the two groups from baseline at 12 month | 1 year
Improvement in liver function test as compared to baseline in both groups. | 1 year
Improvement in HVPG (Hepatic Venous Pressure Gradient) as compared to baseline in both groups. | 1 year
Improvement duodenal biopsy as compared to baseline in both groups. | 1 year
  Improvement is defined as improvement in microbiome pre and post treatment.
Improvement in liver stiffness as measured by fibroscan test as compared to baseline in both groups. | 1 year
Improvement in insulin resistance in both groups. | 1 year
  Improvement is defined as improvement in the fasting plasma and insulin levels, HOMA-IR
Reduction in hepatic and systemic inflammatory markers in both groups | 1 year
  Hepatic and systemic inflammatory like Tumor Necrosis Factor-α, CRP and serum endotoxins.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kapil Dev Jamwal, DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided